CLINICAL TRIAL: NCT00416884
Title: Fludarabine, Campath, TBI T-Cell Deplete NMSCT With Post-Transplant T-Cell Infusions for CML Failing Imatinib Therapy With Imatinib (STI571)
Brief Title: Flu,Alemtuzumab,and TBI Followed By Donor Stem Cell Chronic Phase CML
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Richard Maziarz, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000449649; OHSU-TPI-02032-L (Other: OHSU Knight Cancer Institute); OHSU-414 (Other: OHSU IRB)
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Results first posted 2011-08-02 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2011-07

CONDITIONS: Leukemia
Keywords: chronic phase chronic myelogenous leukemia; childhood chronic myelogenous leukemia; relapsing chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase | interventions — Alemtuzumab; fludarabine; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TBI, Campath, Fludarabine T-cell Deplete (Experimental): (Campath) 30 mg on day -8 over 5-6 hours, Fludarabine 30 mg/m^2 on day -4 through day -2, Total body irradiation single fraction 200 cGy at 7 cGy per minute on day 0., Stem cells will be T cell depleted and given on day 0
  Interventions: Drug: Campath; Drug: Fludarabine; Radiation: Total Body Irradiation (TBI); Other: T-Cell Deplete

INTERVENTIONS:
Drug: Campath — 30 mg on day -8 over 5-6 hours
  Other Names: Nonmeylablative Stem Cell Transplant; Mini Transplant
Drug: Fludarabine — Fludarabine 30 mg/m^2 on day -4 through day -2
  Other Names: Nonmeylablative Stem Cell Transplant; Mini Transplant
Radiation: Total Body Irradiation (TBI) — Total body irradiation single fraction 200 cGy at 7 cGy per minute on day 0
  Other Names: Nonmeylablative Stem Cell Transplant; Mini Transplant
Other: T-Cell Deplete — Stem cells will be T cell depleted and given on day 0
  Other Names: Nonmeylablative Stem Cell Transplant; Mini Transplant

SUMMARY:
RATIONALE: Giving low doses of chemotherapy, such as fludarabine, and total-body irradiation (TBI) before a donor stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune system and help destroy any remaining cancer cells (graft-versus-tumor effect). Giving an infusion of the donor's T cells (donor lymphocyte infusion) that have been treated in the laboratory after the transplant may help increase this effect. Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine and alemtuzumab, and removing the T lymphocyte cells(T cells) from the donor cells before transplant, may stop this from happening.

PURPOSE: This clinical trial is studying how well giving fludarabine, alemtuzumab, and total-body irradiation together with donor stem cell transplant and donor white blood cell (WBC) infusion works in treating patients with chronic phase chronic myelogenous leukemia (CML) that did not respond to previous imatinib mesylate.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the treatment-related mortality in patients with imatinib mesylate-resistant chronic phase chronic myelogenous leukemia treated with nonmyeloablative conditioning comprising fludarabine, alemtuzumab, and total-body irradiation followed by T-cell-depleted allogeneic stem cell transplantation and post-transplantation allogeneic T-cell infusion.
* Determine if donor engraftment can be safely established using partial T-cell depletion with additional T-cell infusions in these patients.

OUTLINE: Patients receive alemtuzumab IV over 5-6 hours on day -8 and fludarabine IV on days -4 to -2. Patients undergo total-body irradiation followed by T-cell-depleted (CD34+ selected) allogeneic stem cell transplantation on day 0. Patients receive allogeneic T-cell infusion on days 30 and 60. Patients also receive cyclosporine twice daily beginning on day -3 and continuing until day 100 followed by a taper until day 177.

PROJECTED ACCRUAL: Not specified.

ELIGIBILITY:
Inclusion criteria:

* Patients aged 4-75 with chronic myelogenous leukemia (CML) treatable by allogeneic hematopoietic stem cell transplant.
* Patients with cytogenetically confirmed chronic phase CML.

  o Hematologic parameters for chronic phase are: i) Percentage of blasts in peripheral blood or marrow < 15% ii) Percentage of blasts + promyelocytes in the peripheral blood or bone marrow < 30% iii) Percentage of basophils in blood or marrow <20% iv) Platelet count > 100 x 109/l
* Patients must have demonstrated refractoriness/resistance to STI571 defined as follows:

  i) Hematologically resistant- failure to achieve a complete hematologic remission (CHR) despite 3 months of STI571 therapy.

ii) Hematologically refractory - a rising WBC count > 20 x 109/l confirmed by two samples taken two weeks apart in a patient with a previous CHR despite concurrent treatment with STI571 iii) Cytogenetically resistant - bone marrow cytogenetics showing > 65% Philadelphia chromosome positivity (Ph+) after 6 months of STI571 based therapy.

iv) Cytogenetically refractory - An increase in the number of Philadelphia chromosome positive (Ph+) bone marrow cells by at least 30%, or an increase to > 65%, confirmed by samples at least 1 month apart following a previous STI571 induced cytogenetic response, while continuing STI571 therapy.

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Patients with a human leukocyte antigen (HLA) matched sibling donor at the HLA-A, B, and DR loci.
* Patients with an unrelated hematopoietic stem cell donor must be matched using high resolution typing for class II human leukocyte antigen (HLA-DR beta-1, 3, 4, 5 and DQ beta-1) and matched with intermediate to high resolution molecular typing at class I human leukocyte antigen (HLA-A, B, and C) loci.
* Patients with accelerated or blast crisis of CML who have returned to chronic phase as described above are eligible.
* Written informed, voluntary consent.

Exclusion criteria:

* Patients who have received another investigational drug within 30 days.
* Fertile men unwilling to use contraceptive techniques during and for 24 months following treatment.
* Females who are pregnant or fertile women unwilling to use contraceptive techniques for two months prior to entering the study and for 24 months following treatment.
* Patients with active bacterial or fungal infections unresponsive to medical therapy.
* Patients with organ dysfunction including cardiac ejection fraction of less than 35% or pulmonary status with a diffusing capacity of the lung for carbon monoxide(DLCO) of less than 40% and/or receiving supplemental oxygen.
* Liver Function Abnormalities: patients will be excluded if they are found to have fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, varices, history of bleeding varices, hepatic encephalopathy or chronic viral hepatitis where the total serum bilirubin is greater than 3 mg per deciliter with symptomatic biliary disease.
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable.
* Patients with a history of any prior bone marrow or peripheral blood stem cell transplantation.
* Patients with any other serious, uncontrolled, concomitant medical condition
* HIV positive patients

Eligibility criteria for donors:

Inclusion Criteria for Donors:

* Sibling donors are permitted if matched at class I human leukocyte antigen (HLA-A, B), and class II human leukocyte antigen (DR) loci.
* Unrelated donors must be matched for class II human leukocyte antigen(HLA-DR beta-1,2,3,4,5) and class II human leukocyte antigen (DQ beta-1) with high resolution typing and with intermediate resolution molecular typing at class I human leukocyte antigen(HLA-A, B, and C) loci.
* Donors must be eligible to serve as a peripheral stem cell allograft donor. Bone marrow donors will not be permitted on this protocol.
* Donors must be >18 and < 75 years of age.

Exclusions Criteria for Donors:

* Volunteer donors who wish to serve as bone marrow donors only and refuse exogenous cytokines.
* Donors who are Human immunodeficiency virus (HIV+), Human T-lymphotropic virus (HTLV-1+), or hepatitis Bs Ag+..
* Donors with medical conditions that would result in increased risk for Granulocyte colony-stimulating factor (G-CSF) mobilization and harvest of peripheral blood stem cells (PBSC) including renal insufficiency with Cr > 2.0, idiopathic splenomegaly, underlying coagulopathy, uncontrolled coronary artery disease, and major surgery within 28 days.

Ages: 4 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2003-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Maziarz, MD, Study Chair — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- TBI, Campath, Fludarabine T-cell Deplete: (Campath) 30 mg on day -8 over 5-6 hours, Fludarabine 30 mg/m2 on day -4 through day -2, Total body irradiation single fraction 200 cGy at 7 cGy per minute on day 0., Stem cells will be T-cell depleted and given on day 0
Period: Overall Study
Arm/Group | TBI, Campath, Fludarabine T-cell Deplete
Started | 1
Completed | 0
Not Completed | 1
Not completed — Study terminated due to low accrual | 1

BASELINE CHARACTERISTICS:
Arm/Group | TBI, Campath, Fludarabine T-cell Deplete
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Mortality
Description: Treatment related mortality is a consequence of both complications of the preparative regimen and systemic immunological rejection which is manifested as graft versus host disease(GVHD). The preparative regimens which include whole body radiation and/or high dose chemotherapy are complicated by single or multi-organ failure and by prolonged myelosuppression that can lead to infections and bleeding
Time Frame: lifetime followup, up to 100 years.
Measure: Number; unit: Participants
Arm/Group | TBI, Campath, Fludarabine T-cell Deplete
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Arm/Group | TBI, Campath, Fludarabine T-cell Deplete
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Study was terminated early due to low enrollment, hence the study did not have any treatment-related mortalities to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No